CLINICAL TRIAL: NCT04485663
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, First-in-human Study of Subcutaneously Administered ALG-010133 to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single Ascending Doses (Part 1) and Multiple Ascending Doses in Healthy Volunteers (Part 2), and Multiple Doses in Subjects With Chronic Hepatitis B (Part 3)
Brief Title: A Study of ALG-010133 Drug to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single and Multiple Doses in Healthy Volunteers and CHB Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of antiviral activity at the projected efficacious dose.
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-010133-101
Record Dates: First submitted 2020-07-09; First posted 2020-07-24 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALG-010133 (Experimental): Subcutaneous injections of ALG-010133 in HV or CHB subjects up to every 7 days for up to 12 weeks
  Interventions: Drug: ALG-010133
- Placebo (Placebo Comparator): Subcutaneous injections of placebo in HV or CHB subjects up to every 7 days for up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALG-010133 — Single or multiple doses of ALG-010133
  Arms: ALG-010133
Drug: Placebo — Single or multiple doses of Placebo
  Arms: Placebo

SUMMARY:
A Randomized Study of ALG-010133 Drug to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single and Multiple Doses in Healthy Volunteers and CHB Subjects

ELIGIBILITY:
Inclusion Criteria for Healthy Subjects:

1. Male and Female between 18 and 55 years old
2. Female subjects must have a negative serum pregnancy test at screening
3. Subjects must be nonsmokers for at least 3 months prior to randomization
4. BMI 18.0 to 32.0 kg/m^2
5. Subjects must have a 12-lead ECG that meets protocol criteria

Inclusion Criteria for CHB Subjects:

1. Male and Female between 18 and 70 years old
2. Female subjects must have a negative serum pregnancy test at screening
3. BMI 18.0 to 35.0 kg/m^2
4. HBeAg-negative chronic hepatitis B or HBeAg-positive chronic hepatitis B and are currently receiving HBV NA treatment for ≥6 months prior to screening
5. Subjects must have a 12-lead ECG that meets protocol criteria

Exclusion Criteria for Healthy Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subject with current or history of clinically significant (as determined by the Investigator) skin disease requiring intermittent or chronic treatment
5. Excessive use of alcohol defined as regular consumption of ≥14 units/week for women and ≥21 units/week for men
6. Unwilling to abstain from alcohol use for 48 hours prior to start of dosing through end of study follow up
7. Subjects with Hepatitis A, B, C, D, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
8. Subjects with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m^2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)

Exclusion Criteria for CHB Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subject with current or history of clinically significant (as determined by the Investigator) skin disease requiring intermittent or chronic treatment
5. Excessive use of alcohol defined as regular consumption of ≥14 units/week for women and ≥21 units/week for men
6. Subjects with Hepatitis A, C, D, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
7. Subjects with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m^2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
8. Subject with any history or current evidence of hepatic decompensation such as: variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy, or active jaundice (within the last year)
9. Subjects must have absence of signs of hepatocellular carcinoma
10. Subjects with history or current liver cirrhosis
11. Subjects positive for anti-HBs anitbodies
12. Subjects with liver fibrosis that is classified as Metavir Score ≥F3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 15 days for Part 1
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 29 days for Part 2
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 162 days for Part 3
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Predose (0 hours) up to 162 Days (3864 hours)
  Pharmacokinetic parameters of ALG-010133 in plasma
Area under the concentration time curve [AUC] | Predose (0 hours) up to 162 Days (3864 hours)
  Pharmacokinetic parameters of ALG-010133 in plasma
Time to maximum plasma concentration [Tmax] | Predose (0 hours) up to 162 Days (3864 hours)
  Pharmacokinetic parameters of ALG-010133 in plasma
Half-time [t1/2] | Predose (0 hours) up to 162 Days (3864 hours)
  Pharmacokinetic parameters of ALG-010133 in plasma
Minimum Plasma Concentration [Cmin] | Predose (0 hours) up to 162 Days (3864 hours)
  Pharmacokinetic parameters of ALG-010133 in plasma
Change in HBsAg (reduction) from baseline through Day 78 in Multiple Dose HBV Infected Patients | Screening, Day -1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78

CONTACTS AND LOCATIONS:
Locations (10):
- China (2):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Jilin University, Changchun, Jilin
- Queen Mary Hospital, Hong Kong, Hong Kong
- PMSI Republican Clinical Hospital "T. Mosneaga", ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- ACS, Auckland, New Zealand
- South Korea (4):
  - Pusan National University Hospital, Busan
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- King's College Hospital, London, United Kingdom